CLINICAL TRIAL: NCT04368195
Title: Evaluation of Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Sleeve Gastrectomy: A Prospective, Randomized, Controlled Clinical Trial
Acronym: ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Consultant Anaesthetist, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-01-R-069
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: Erector spinae block; Upper GI laparoscopy; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group will not receive any regional block
- Erector spinae block group (Experimental): This group will receive erector spinae block
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: Erector spinae block — Erector Spinae Plane Block (ESPB) - first recently described for the treatment of thoracic neuropathic pain, is a peri-paravertebral regional anesthesia technique that has since been reported as an effective technique for prevention of postoperative pain in various surgeries (10-12). In ESPB, local anesthetic is reported to be administered in to the interfascial plane between the transverse process of the vertebra and the erector spinae muscles, spreading to multiple paravertebral spaces.
  Arms: Erector spinae block group

SUMMARY:
This study will help us in understanding the role of erector spinae block (ESPB) for postoperative pain control in patients undergoing upper GI laparoscopy surgeries. The surgeries included in this group include laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic umblical or epigastric hernia repair. Patients aged between 18 and 65 years, scheduled to undergo any upper GI laparoscopy surgeries with an ASA score of 1 or 2 will be included in the study. This is a prospective randomised controlled trial which will compare two groups receiving either erector spinae block or no block for postoperative pain control after upper GI laparoscopy surgeries

DETAILED DESCRIPTION:
Research Proposal and significance Postoperative analgesia should include strategies to reduce side effects. Intravenous analgesics are generally considered to be adequate for pain management in upper GI laparoscopic surgeries. However opioids can lead to nausea, vomiting and itching while NSAIDs affect the gastric, hepatic and renal systems and wound healing. Reducing opioid requirements during the perioperative period is among the current goals of enhanced recovery programs. The objective is to reduce all potential opioid-related side-eﬀects. Therefore, multimodal analgesics including regional blocks decrease the use of other analgesics and therefore decrease side effects.

Objective The aim of this study is to evaluate the eﬀect of Erector spinae block (ESPB) on postoperative pain in upper GI laparoscopy surgeries, which leads to both visceral and somatic pain.

Research review In this study, the surgeries included in upper GI laparoscopic surgeries are laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic umblical or epigastric hernia repair.

n upper GI laparoscopy surgeries, postoperative pain is caused by two reasons; one is somatic pain from the trocar entry incisions and additionally peritoneal distention and diaphragm irritation due to high intra-abdominal pressure and CO2 insufflations lead to visceral pain as well. Therefore, any analgesic protocol for these surgeries must be effective on both sources of pain.

Regional block techniques studied and considered part of multimodal anesthesia include transversus abdominis plane block (TAP), oblique subcostal transversus abdominis plane block (OSTAP or STAP) and paravertebral block. Apart from paravertebral block, these techniques only effect somatic pain and can therefore be inadequate in some cases. Ultrasound Guided paravertebral block is an advanced regional anesthesia technique. When considering that the pleura forms one boundary of the paravertebral space, ESPB can be considered an easier technique to perform. It is also safer because the needle remains behind the transverse process. However, non-inferiority studies comparing ESPB and paravertebral block are required. Erector Spinae Plane Block (ESPB) - first recently described for the treatment of thoracic neuropathic pain, is a peri-paravertebral regional anesthesia technique that has since been reported as an effective technique for prevention of postoperative pain in various surgeries. In ESPB, local anesthetic is reported to be administered in to the interfascial plane between the transverse process of the vertebra and the erector spinae muscles, spreading to multiple paravertebral spaces. Case reports have reported that ESPB effects both the ventral and dorsal rami and leading to blockage of both visceral and somatic pain. Anatomical dissection indicates that the likely mechanism of action is diffusion of local anaesthetic anteriorly through the connective tissues and ligaments spanning the adjacent transverse processes and into the vicinity of the spinal nerve roots. This is consistent with other reports of successful analgesia following injection into a similar tissue plane in the thorax.

Tulgara et al in their study has shown that ultrasound guided bilateral single shot ESPB performed before general anesthesia induction in LC patients signiﬁcantly lowered NRS at rest in the ﬁrst 3h and lead to less analgesia requirement in the ﬁrst 24h when compared to a control group.

Methodology Patients aged between 18 and 65years, scheduled to undergo any upper GI laparoscopy surgeries with an ASA score of 1 or 2 will be included in the study. Written informed consent for general anesthesia and all procedures will be obtained from all patients. Patients who refused enrollment or later requested removal for the study, those who are unable to give informed consent and patients with either contraindications for regional anesthesia, known allergy to local anesthetics, bleeding diathesis, use of anticoagulants or corticosteroids, inability to operate patient controlled analgesia (PCA) system, psychiatric disorders or use of psychiatric medications and conversion to open laparotomy will not be included in the study.

There will be two groups of patients: control group (Group A) and ESPB group (Group B). Upon ward admission, a random ID will assigned to each patient. Simple randomization in the operating room will performed using the closed envelope method to determine which group the patient would be included in.

The random ID assigned to each patient will be used when collecting all patient data in the ward postoperatively. The anesthesiologist performing the simple randomization will also perform the block but will not play any role in the collection of postoperative data or its analysis.

General anesthesia and surgical technique will be the same for both groups. Standard monitoring procedures included pulse oximetry, electrocardiography, and noninvasive arterial pressure will be performed prior to anesthesia. Baseline heart rates, systolic and diastolic blood pressures, and mean arterial pressures will be recorded before anesthesia. Induction will performed using propofol 2-3 mgkg-1, fentanyl 100μg and Cisatracurium 0.2 mgkg-1. 0.8-1.0 MAC sevoﬂurane and 0.05-0.1 μg/kg/min remifentanil infusion will be used for anesthesia maintenance. Remifentanil dosage will be adjusted according to hemodynamic parameters, up to 2 μg/kg/min. Standard perioperative intravenous analgesia protocol will include paracetamol 1g and Lornoxicam 16 mg.After completion of surgery, patients will be extubated once TOF ratio of >0.9 is acheived and transferred to the recovery room. Local anesthesia will not be applied to wounds. Pneumoperitoneum will be evacuated in all patients at the end of surgery. All patients will receive 8 mg Dexamethasone and 1 mg Granisteron as antiemtics.

All blocks will be performed in lateral position after general anesthesia induction. ESPB will be performed under ultrasonographic guidance using a linear 6- to 10-MHz ultrasound probe. The linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3cm lateral to the T9 spinous process. The erector spinae muscles will be identiﬁed superﬁcial to the tip of the T9 transverse process. A 21-gauge 10-cm needle will be inserted using an in-plane superior-to-inferior approach or an outplane approach. The tip of the needle will be placed into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will conﬁrmed by visible ﬂuid spread lifting erector spinae muscle oﬀ the bony shadow of the transverse process on ultrasonographic imaging. A total of 10-15 mL of 0.2% ropivacaine will be injected each side.

The Numeric Rating Scale (NRS) will be used to evaluate postoperative pain. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reﬂects the intensity of his/her pain. It is considered a one dimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme ("no pain") to'10' representing the other pain extreme ("pain as bad as you can imagine" or "worst pain imaginable"). Changes in NRS at rest and on movement will be recorded at intervals.

All patients will be followed using a standardized postoperative analgesia protocol which includes Morphine PCA. Morphine at a concentration of 1mg/ml is included in our PCA protocol (total volume 100mL.) PCAs will be set as no basal infusion and 1 mg bolus doses with a 10 min lock out time. PCA will be commenced when the patient arrives in the recovery room. For rescue analgesia during the ﬁrst hour in the recovery room, 2 mg Morphine will be used if NRS≥4/10. The dosage will be repeated every 20 min if NRS > 4/10. Paracetamol 1g / 8h will be used during ward follow-up. If NRS < 2 and the patient refuses pain medication, this dosage will be skipped. As rescue analgesia in case of the pain score≥4/10 on NRS during 1-24h, Lornoxicam 16 mg IV will be performed. If the pain remains at same level in following 1h period Morphine 2 mg IV will be added. Patient will receive 1 mg Granisetron IV if complains of nausea/vomiting.

Primary outcome measures at commencement of the study will be NRS pain score at 18th hours postoperatively both at rest and when coughing. Secondary outcome measures will be routine (paracetamol or morphine PCA) or rescue analgesic use within the ﬁrst 24h. In addition to the above measures, NRS pain scores will measured at other time intervals like 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours and 24 hours postoperatively. Also, shoulder pain during the ﬁrst 24 h and presence of postoperative nausea and vomiting will be noted. The severity of both nausea and sedation will be assessed by patients on a 4 point scale (none, mild, moderate, and severe). Nurses will note any vomiting in the recovery room or on the ward. Finally, the number of patients receiving Granisetron will be recorded.

The null hypothesis of our study is that there is no diﬀerence in pain scores between ESPB and a control group receving standard analgesic regimen in patients undergoing upper GI laparoscopic surgeries.

For sample size calculation, we used the study by Tulgara et al (16) done on laparoscopic cholecystectomy with pooled standard deviation of 0.725 and margin of error (d) as 0.6 units on NRS scale at α=0.05 and power 80 %.

The sample size was calculated using the formula n = 2 ( Zα + Zβ) 2 X σ2/d2

where Zα = 1.96 ( 95% confidence interval), Zβ = 0.84 ( 80% power), σ = 0.725, d = 0.6 Sample size calculated from this formula came out to be 22 in each group and with 10 % dropouts/attrition, it was 25 patients in each group.

SPSS 16.0 Statistical package programme (SPSS, Chicago, IL, USA) will be used for statistical analysis. Descriptive statistics will be expressed as mean ± standard deviation. Univariate analysis compare in groups means using a 2-sample, independent t-test assuming equal variances for continuous variables. For data without normal distribution, Mann Whitney U test will be performed. Ratios will be compared using Chi-Square. Categorical variables will be compared using Fisher exact test. A p-value of<0.05 is considered statistically signiﬁcant. NRS will be analysed using repeated measures analysis.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65years, scheduled to undergo any upper GI laparoscopy surgeries with an ASA score of 1 or 2 will be included in the study. The surgeries included in this group include laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic umblical or epigastric hernia repair.

Written informed consent for general anesthesia and all procedures will be obtained from all patients.

Exclusion Criteria:

* Patients who refused enrollment or later requested removal for the study, those who are unable to give informed consent and patients with either contraindications for regional anesthesia, known allergy to local anesthetics, bleeding diathesis, use of anticoagulants or corticosteroids, inability to operate patient controlled analgesia (PCA) system, psychiatric disorders or use of psychiatric medications and conversion to open laparotomy will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
NRS pain score at 18th hours | 18th hour
  Primary outcome measures at commencement of the study will be NRS pain score at 18th hours postoperatively both at rest and when coughing.

SECONDARY OUTCOMES:
Analgesic consumption | 24 hours
  Secondary outcome measures will be routine (paracetamol or morphine PCA) or rescue analgesic use within the ﬁrst 24h.
Adverse events | 24 hours
  Adverse events like shoulder pain during the ﬁrst 24 h and presence of postoperative nausea and vomiting will be noted. The severity of both nausea and sedation will be assessed by patients on a 4 point scale (none, mild, moderate, and severe).

OTHER OUTCOMES:
NRS pain score at other time intervals | 0-24 hours
  NRS pain scores will also be measured at 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours and 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Security Forces Hospital Program, Riyadh
  - Security Forces Hospital, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year

REFERENCES:
- [Result] Adhikary SD, Bernard S, Lopez H, Chin KJ. Erector Spinae Plane Block Versus Retrolaminar Block: A Magnetic Resonance Imaging and Anatomical Study. Reg Anesth Pain Med. 2018 Oct;43(7):756-762. doi: 10.1097/AAP.0000000000000798. PMID 29794943
- [Result] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Result] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Result] Singla S, Mittal G, Raghav, Mittal RK. Pain management after laparoscopic cholecystectomy-a randomized prospective trial of low pressure and standard pressure pneumoperitoneum. J Clin Diagn Res. 2014 Feb;8(2):92-4. doi: 10.7860/JCDR/2014/7782.4017. Epub 2014 Feb 3. PMID 24701492
- [Result] Enes H, Semir I, Sefik H, Husnija M, Goran I. Postoperative pain in open vs. laparoscopic cholecystectomy with and without local application of anaesthetic. Med Glas (Zenica). 2011 Aug;8(2):243-8. PMID 21849946
- [Result] Shin HJ, Oh AY, Baik JS, Kim JH, Han SH, Hwang JW. Ultrasound-guided oblique subcostal transversus abdominis plane block for analgesia after laparoscopic cholecystectomy: a randomized, controlled, observer-blinded study. Minerva Anestesiol. 2014 Feb;80(2):185-93. Epub 2013 Oct 31. PMID 24193176
- [Result] Oksar M, Koyuncu O, Turhanoglu S, Temiz M, Oran MC. Transversus abdominis plane block as a component of multimodal analgesia for laparoscopic cholecystectomy. J Clin Anesth. 2016 Nov;34:72-8. doi: 10.1016/j.jclinane.2016.03.033. Epub 2016 May 2. PMID 27687350
- [Result] Visoiu M, Cassara A, Yang CI. Bilateral Paravertebral Blockade (T7-10) Versus Incisional Local Anesthetic Administration for Pediatric Laparoscopic Cholecystectomy: A Prospective, Randomized Clinical Study. Anesth Analg. 2015 May;120(5):1106-1113. doi: 10.1213/ANE.0000000000000545. PMID 25427288
- [Result] Petersen PL, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB, Mathiesen O. The beneficial effect of transversus abdominis plane block after laparoscopic cholecystectomy in day-case surgery: a randomized clinical trial. Anesth Analg. 2012 Sep;115(3):527-33. doi: 10.1213/ANE.0b013e318261f16e. Epub 2012 Jul 4. PMID 22763903
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Aksu C, Gurkan Y. Ultrasound guided erector spinae block for postoperative analgesia in pediatric nephrectomy surgeries. J Clin Anesth. 2018 Mar;45:35-36. doi: 10.1016/j.jclinane.2017.12.021. Epub 2017 Dec 20. No abstract available. PMID 29274546
- [Result] Balaban O, Aydin T, Yaman M. Is ultrasound guided erector spinae plane block sufficient for surgical anesthesia in minor surgery at thoracal region? J Clin Anesth. 2018 Jun;47:7-8. doi: 10.1016/j.jclinane.2018.02.012. Epub 2018 Mar 6. No abstract available. PMID 29522967
- [Result] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Result] Restrepo-Garces CE, Chin KJ, Suarez P, Diaz A. Bilateral Continuous Erector Spinae Plane Block Contributes to Effective Postoperative Analgesia After Major Open Abdominal Surgery: A Case Report. A A Case Rep. 2017 Dec 1;9(11):319-321. doi: 10.1213/XAA.0000000000000605. PMID 28727597
- [Result] Costache I, Sinclair J, Farrash FA, Nguyen TB, McCartney CJ, Ramnanan CJ, Goodwin SL. Does paravertebral block require access to the paravertebral space? Anaesthesia. 2016 Jul;71(7):858-9. doi: 10.1111/anae.13527. No abstract available. PMID 27291614
- [Result] Roue C, Wallaert M, Kacha M, Havet E. Intercostal/paraspinal nerve block for thoracic surgery. Anaesthesia. 2016 Jan;71(1):112-3. doi: 10.1111/anae.13358. No abstract available. PMID 26684531
- [Result] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Derived] Ul Huda A, Alshahrani AS, Yasir M, Sawilah A, Alharthi AAN. Erector spinae block reduces intraoperative and postoperative opioid consumption in patients undergoing laparoscopic sleeve gastrectomy: A randomized controlled trial. Qatar Med J. 2024 Dec 26;2024(4):58. doi: 10.5339/qmj.2024.58. eCollection 2024. PMID 39944209